CLINICAL TRIAL: NCT02812576
Title: Burden of Invasive Group B Streptococcal Disease in Infants and Resistance Surveillance in China---A National, Multi-center, Prospective Observational Study
Brief Title: Burden of Invasive Group B Streptococcal Disease in Infants and Resistance Surveillance in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xi'an Jiaotong University (Other)
Collaborators: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Haiying Liu, Director of Clinical Laboratory, Guangzhou Women and Children's Medical Center
Other Study IDs: XJTU-CDSP_01
Record Dates: First submitted 2016-06-13; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Invasive Group B Streptococcal Disease
Keywords: Group B streptococcus; Infants; China

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Data on neonatal GBS disease are very limited in China. Acceptance and implementation of prevention measures such as antibiotics prevention or vaccination against GBS disease would require robust data. This study as the first national, multicenter study to investigate the epidemiology of GBS disease in China, and the resistance surveillance of GBS isolates, to appraise the necessity of appropriate interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Positive culture for GBS from normally sterile sites such as blood or cerebrospinal fluid.
2. ≤90 days old at the time of GBS confirmation.
3. Voluntary written informed consent provided.

Exclusion Criteria:

1. None

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants <3 months old born in or treated in a study hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of group B streptococcal (GBS) disease | From birth to 3 months of age
Case Fatality Rate of GBS disease | From birth to 3 months of age
GBS serotype distribution | From birth to 3 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Haiying Liu, MD, Ph.D, Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (1):
- Health Science Center of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ji W, Zhou H, Li J, Britto CD, Liu Z, Zhang W, Du J, Madhi SA, Kwatra G, Dangor Z, Jin Z, Zhao H, Zhao Y, Fang Y, Li J. Distributions of candidate vaccine Targets, virulence Factors, and resistance features of invasive group B Streptococcus using Whole-Genome Sequencing: A Multicenter, population-based surveillance study. Vaccine. 2024 Jun 11;42(16):3564-3571. doi: 10.1016/j.vaccine.2024.04.062. Epub 2024 Apr 30. PMID 38692955
- [Derived] Ji W, Liu H, Jin Z, Wang A, Mu X, Qin X, Wang W, Gao C, Zhu Y, Feng X, Lei J, She S, Jiang L, Liu J, Yang S, Liu Z, Li G, Li Q, Guo D, Aziz MM, Gillani AH, Fang Y. Disease burden and antimicrobial resistance of invasive group B streptococcus among infants in China: a protocol for a national prospective observational study. BMC Infect Dis. 2017 May 31;17(1):377. doi: 10.1186/s12879-017-2475-9. PMID 28569141